CLINICAL TRIAL: NCT04114643
Title: Prothrombin Complex Concentrate Versus Frozen Plasma in Bleeding Adult Cardiac Surgical Patients: A Multicentre, Randomized, Active-control, Pragmatic, Phase 2 Pilot Study
Brief Title: Factor Replacement in Surgery
Acronym: FARES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-5393
Record Dates: First submitted 2019-09-25; First posted 2019-10-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-07

CONDITIONS: Bleeding in Cardiac Surgery
Keywords: Frozen Plasma (FP); Prothrombin Complex Concentrate (PCC); Octaplex; Coagulation Factor Replacement; Transfusion; Bleeding Cardiac Surgical Patients; Pilot; Phase 2
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX; prothrombin complex concentrates

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either PCC or FP when the blood bank receives the first order for coagulation factor replacement and deems it to be in accordance with accepted clinical standards.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prothrombin Complex Concentrate (Active Comparator)
  Interventions: Biological: Prothrombin Complex Concentrate
- Frozen Plasma (Active Comparator)
  Interventions: Biological: Frozen Plasma

INTERVENTIONS:
Biological: Prothrombin Complex Concentrate — Octaplex will be administered when the blood bank receives an order for coagulation factor replacement
  Other Names: Octaplex
  Arms: Prothrombin Complex Concentrate
Biological: Frozen Plasma — Frozen Plasma will be administered when the blood bank receives an order for coagulation factor replacement
  Other Names: Fresh Frozen Plasma
  Arms: Frozen Plasma

SUMMARY:
This is a multicentre, randomized, active-control, pragmatic, Phase 2 pilot study in adult cardiac surgery patients. Two Canadian hospitals will participate, and it is estimated that the study will take approximately 9 months to complete.

Approximately 120 bleeding adult cardiac surgical patients who require coagulation factor replacement during cardiac surgery will be included. Patients will be randomized to receive either PCC or FP when the blood bank receives the first order for coagulation factor replacement and deems it to be in accordance with accepted clinical standards. Patients will be treated according to their assigned group on the first and second times when coagulation factor replacement is ordered during the treatment period (24 hours after randomization). For any additional doses (i.e., the third dose and thereafter), patients in both groups will receive FP (in 1U increments at the discretion of the ordering physician). No other aspects of care will be modified.

This pilot study aims to select a clinically relevant primary efficacy endpoint for a confirmative Phase 3 study, which will subsequently aim to determine if PCC is non-inferior or superior to FP in terms of effica-cy and safety in bleeding cardiac surgical patients. In the pilot study, safety outcomes will be measured for the first 28 days, which is the duration of participation of each patient in the trial.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing any index cardiac surgery with or without CPB in whom coagulation factor replacement with PCC or FP is ordered in the operating room for:

1. Management of bleeding, or
2. Anticipated bleeding in a patient who has

   1. been on-pump for >2 hours, or
   2. undergone a complex procedure (e.g., ACB + AVR). Coagulation factor deficiency must either be known to exist (as indicated by elevated EXTEM clotting time [CT] or international normalized ratio [INR]), or be suspected based on the clinical situation.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

1. Undergoing heart transplantation, insertion or removal of ventricular assist devices (not including intra-aortic balloon pump [IABP]), or repair of thoracoabdominal aneurysm
2. Critical state immediately before emergency surgery with high probability of death within 24 hours of surgery (e.g., acute aortic dissection, cardiac arrest within 24 hours before start of surgery)
3. History of heparin induced thrombocytopenia
4. Last preoperative INR >1.5 and patient on warfarin
5. Taken dabigatran, rivaroxaban, apixaban, or edoxaban within 48 hours of start of surgery
6. Administered PCC or FP within 48 hours before start of surgery
7. History of severe allergic reaction to PCC or FP
8. Refusal of allogeneic blood products due to religious or other reasons
9. Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response | At 4 and 24 hours
  Administration of hemostatic agents including a second dose of IMP, platelet transfusion, or surgical re-exploration
Amount of allogeneic blood products | 24 hours after the start of surgery
Number of patients who do not receive any RBC transfusions or any allogeneic blood transfusions | first 24 hours after the start of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Karkouti, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayes K, Fernando MC, Jordan V. Prothrombin complex concentrate in cardiac surgery for the treatment of coagulopathic bleeding. Cochrane Database Syst Rev. 2022 Nov 21;11(11):CD013551. doi: 10.1002/14651858.CD013551.pub2. PMID 36408876
- [Derived] Karkouti K, Bartoszko J, Grewal D, Bingley C, Armali C, Carroll J, Hucke HP, Kron A, McCluskey SA, Rao V, Callum J. Comparison of 4-Factor Prothrombin Complex Concentrate With Frozen Plasma for Management of Hemorrhage During and After Cardiac Surgery: A Randomized Pilot Trial. JAMA Netw Open. 2021 Apr 1;4(4):e213936. doi: 10.1001/jamanetworkopen.2021.3936. PMID 33792729